CLINICAL TRIAL: NCT03552289
Title: Randomized Clinical Study to Evaluate the Advance® Enforcer™ 35 Focal-Force PTA Balloon Catheter in Treatment of Arteriovenous Dialysis Access Circuit Stenosis
Brief Title: Cook Enforcer Post-Market Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-04
Record Dates: First submitted 2018-05-17; First posted 2018-06-11 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: End-Stage Renal Disease
Keywords: Dialysis; Renal; Hemodialysis; Stenosis(es); Transluminal; Percutaneous Transluminal Angioplasty
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cook Enforcer balloon catheter (Active Comparator): The Enforcer balloon will be used in the treatment of obstructive lesions of native or synthetic arteriovenous dialysis fistula.
  Interventions: Device: Cook Advance® Enforcer 35 Focal-Force Percutaneous Transluminal Angioplasty (PTA) Balloon Catheter
- Conventional angioplasty balloon catheters (Active Comparator): Commercially available angioplasty balloon devices will be used in the treatment of obstructive lesions of native or synthetic arteriovenous dialysis fistula.
  Interventions: Device: Conventional angioplasty balloon catheters

INTERVENTIONS:
Device: Cook Advance® Enforcer 35 Focal-Force Percutaneous Transluminal Angioplasty (PTA) Balloon Catheter — The Enforcer balloon device will be used in treatment of obstructive lesions of native or synthetic arteriovenous dialysis fistula
  Arms: Cook Enforcer balloon catheter
Device: Conventional angioplasty balloon catheters — Commercially available angioplasty balloon devices will be used in treatment of obstructive lesions of native or synthetic arteriovenous dialysis fistula
  Arms: Conventional angioplasty balloon catheters

SUMMARY:
The purpose of this study is to evaluate the performance of the Cook Advance® Enforcer™ 35 Focal-Force PTA Balloon Catheter (or Enforcer balloon) in treating narrowed blood vessels compared to treatment with a conventional angioplasty balloon.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or physiological abnormalities which indicate dialysis access dysfunction (e.g., decreased access blood flow, elevated venous pressure, decreased dialysis dose, abnormal physical exam)

Exclusion Criteria:

* Less than 18 years old
* Pregnant, lactating, or planning to become pregnant in the 3 months following enrollment
* Underwent any surgical or interventional procedure of the access circuit less than or equal to 30 days prior to enrollment
* Scheduled for a kidney transplant
* Stent or stent graft in the arteriovenous (AV) dialysis access circuit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arizona Kideny Disease & Hypertension Surgery Center, Phoenix, Arizona
  - The Vascular Experts, Darien, Connecticut
  - Delaware Kidney/Nephrology Associates, PA, Newark, Delaware
  - Fairlawn Surgery Center, Roanoke, Virginia
  - Vascular Institute of Virginia, Woodbridge, Virginia

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Lesions
Groups:
- Conventional Angioplasty Balloon Catheters: Commercial available angioplasty balloon devices will be used in the treatment of obstructive lesions of native or synthetic arteriovenous dialysis fistula.
  Conventional angioplasty balloon catheters: Commercial available angioplasty balloon devices will be used in treatment of obstructive lesions of native or synthetic arteriovenous dialysis fistula
Period: Overall Study
Arm/Group | Cook Enforcer Balloon Catheter | Conventional Angioplasty Balloon Catheters
Started | 102; 120 Lesions | 109; 130 Lesions
Completed | 101; 119 Lesions | 106; 125 Lesions
Not Completed | 1; 1 Lesions | 3; 5 Lesions

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cook Enforcer Balloon Catheter | Conventional Angioplasty Balloon Catheters | Total
Number analyzed (Participants) | 102 | 109 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (12.4) | 65.5 (12.8) | 65.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 51 | 94
  Male | 59 | 58 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 15 | 20
  Not Hispanic or Latino | 97 | 93 | 190
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 43 | 86
  White | 51 | 57 | 108
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 7 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent of Lesions Requiring Adjunctive Treatment
Description: Percentage of lesions requiring adjunctive treatment immediately following the initial treatment with the Enforcer or conventional angioplasty balloon
Time Frame: Immediately following treatment of stenoses of a mature native arteriovenous dialysis access circuit fistula or graft, up to approximately 1 hour
Measure: Count of Units; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Cook Enforcer Balloon Catheter | Conventional Angioplasty Balloon Catheters
Number analyzed (Participants) | 102 | 109
Number analyzed (Lesions) | 120 | 130
Lesions | 30 | 26
Statistical Analysis 1: Comparison: Cook Enforcer Balloon Catheter vs Conventional Angioplasty Balloon Catheters; Test type: Superiority; p = 0.8283, One-sided Z-test

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Cook Enforcer Balloon Catheter | Conventional Angioplasty Balloon Catheters
All-Cause Mortality (participants affected / at risk) | 1/102 | 2/109
Serious Adverse Events (participants affected / at risk) | 2/102 | 1/109
Other Adverse Events (participants affected / at risk) | 24/102 | 23/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cook Enforcer Balloon Catheter (N=102) | Conventional Angioplasty Balloon Catheters (N=109)
Right Femur Fracture after fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic ulcer of lower extremity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Head injury s/p fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cook Enforcer Balloon Catheter (N=102) | Conventional Angioplasty Balloon Catheters (N=109)
Restenosis or occlusion (Vascular disorders) | 24 (26) | 19 (23)
Thrombosis (Vascular disorders) | 2 (3) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT03552289/Prot_SAP_000.pdf